CLINICAL TRIAL: NCT04638660
Title: Randomized, Placebo-Controlled, Double-Masked Study of the Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) in Subjects With Dim Light Vision Disturbances
Brief Title: Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) in Subjects With Dim Light Vision Disturbances
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXDLD-301 (LYNX-1)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2023-08

CONDITIONS: Dim Light Vision Disturbances
Keywords: Nyxol, Night Vision Disturbances, Glare, Halos, Starbursts

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized into the study in a 1:1 ratio to one of the treatment arms (Nyxol or placebo), with a stratification by light/dark irides.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Ophthalmic Solution 0.75% (Experimental): One drop in both eyes at or near bedtime (8PM to 10PM)
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%
- Phentolamine Ophthalmic Solution Vehicle (Placebo Comparator): One drop in both eyes at or near bedtime (8PM to 10PM)
  Interventions: Drug: Phentolamine Ophthalmic Solution Vehicle (Placebo)

INTERVENTIONS:
Drug: Phentolamine Ophthalmic Solution 0.75% — 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol; Nyxol®
  Arms: Phentolamine Ophthalmic Solution 0.75%
Drug: Phentolamine Ophthalmic Solution Vehicle (Placebo) — Topical sterile ophthalmic solution
  Arms: Phentolamine Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of Nyxol to improve mesopic low contrast visual acuity (mLCVA) in subjects with Dim Light Vision Disturbances (DLD)
* To evaluate efficacy of Nyxol to improve visual performance
* To evaluate the safety of Nyxol

DETAILED DESCRIPTION:
Placebo-controlled, double-masked, multiple-dose, Phase 3 study in approximately 160 randomized subjects with DLD (approximately 136 that are evaluable for efficacy), evaluating safety and efficacy of Nyxol in subjects with DLD following administration of Nyxol once daily (QD) at or near bedtime (at 8PM to 10PM) in both eyes (OU) for 14 days.

Following the successful completion of screening, each subject will be stratified by iris color (light/dark irides) and will then be randomized to treatment (masked) 1:1, Nyxol or placebo (vehicle).

Treatment (Nyxol or placebo) will be administered in both eyes (OU) by the subjects at or near bedtime each day.

At the first visit subjects will be screened for study eligibility.

Treatment visits will occur 2 times: Day 8 (+1 day)/Visit 2 and Day 15 (+1 day)/Visit 3. mLCVA evaluations shall be performed on each of these days.

A follow-up visit (Visit 4) phone call will occur 1 to 3 days after Visit 3.

At select sites OPD Scan measurements will be made using wavefront abhermettry.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Subject-reported DLD (likely subjects with a history of multifocal IOLs, post-laser-assisted in situ keratomileusis [LASIK], corneal scars, and keratoconus)
3. Ability to comply with all protocol-mandated procedures independently and to attend all
4. Otherwise healthy and well-controlled subjects
5. Able and willing to give written consent to participate in this study
6. Able to self-administer study medication
7. PD ≥ 6 mm under mesopic conditions (prior to illumination) in at least one eye
8. ≤ 20 (20/100 Snellen or worse) ETDRS letters in mLCVA score
9. ≥10 ETDRS letters ( ≥2 lines) improvement in mLCVA in at least one eye during illumination of the contralateral eye with a BAT system on low setting

Exclusion Criteria:

Ophthalmic:

1. Prior history of dry eye diagnosis, taking prescription drops for dry eye, or taking artificial tear drops occasionally for dry eye
2. Prior history of fluctuating vision
3. Clinically significant ocular disease as deemed by the Investigator that might interfere with the study
4. Known hypersensitivity to any topical alpha-adrenoceptor antagonists
5. Known allergy or contraindication to any component of the vehicle formulation
6. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal
7. Ocular trauma, ocular surgery (e.g., IOLs) or laser procedure (e.g., LASIK, photorefractive keratectomy [PRK]) within 6 months prior to screening
8. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind within 7 days of screening
9. Recent or current evidence of ocular infection or inflammation in either eye. Subjects must be symptom free for at least 7 days.
10. History of diabetic retinopathy, diabetic macular edema, or dry or wet macular degeneration
11. History of any traumatic (surgical or nonsurgical) or nontraumatic condition affecting the pupil or iris
12. Unwilling or unable to discontinue use of contact lenses at screening until study completion, except for keratoconus subjects who may wear contacts up to 24 hours prior to their scheduled visits

Systemic:

1. Known hypersensitivity or contraindication to alpha- and/or beta-adrenoceptor antagonists
2. Clinically significant systemic disease that might interfere with the study
3. Initiation of treatment with or any changes to the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to screening or during the study
4. Participation in any investigational study within 30 days prior to screening and during the conduct of the study
5. Females of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control
6. Resting HR outside the specified range (50-110 beats per minute)
7. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Clinical Site 6, Newport Beach, California
  - Clinical Site 1, Petaluma, California
  - Clinical Site 3, Jacksonville, Florida
  - Clinical Site 18, Jacksonville, Florida
  - Clinical Site 13, Pittsburg, Kansas
  - Clinical Site 20, Edgewood, Kentucky
  - Clinical Site 14, Louisville, Kentucky
  - Clinical Site 10, Palisades Park, New Jersey
  - Clinical Site 8, Pennington, New Jersey
  - Clinical Site 4, Elizabeth City, North Carolina
  - Clinical Site 22, High Point, North Carolina
  - Clinical Site 9, High Point, North Carolina
  - Clinical Site 2, Fargo, North Dakota
  - Clinical Test 15, Warwick, Rhode Island
  - Clinical Site 11, Memphis, Tennessee
  - Clinical Site 5, San Antonio, Texas
  - Clinical Site 19, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Started | 71 | 73
Completed | 68 | 73
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 70 | 73 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14.14) | 45.4 (14.40) | 46.2 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 120
  Male | 9 | 14 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 66 | 64 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 73 | 143

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With 3 Lines mLCVA Improvement in Study Eye
Description: Percent of subjects with ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (≥3 lines) of improvement in the study eye compared to baseline in monocular mLCVA at Day 8
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Groups:
- Phentolamine Ophthalmic Solution Vehicle: One drop in both eyes at or near bedtime (8PM to 10PM)
  Phentolamine Ophthalmic Solution Vehicle (Placebo): Topical sterile ophthalmic solution Phentolamine Ophthalmic Solution Vehicle
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 70 | 73
Participants | 9 | 2

2. Secondary Outcome: Percent of Subjects With mLCVA Improvement in Study Eye
Description: Percent of subjects with ≥ 5, ≥ 10, and ≥ 15 ETDRS letters (≥ 1, ≥ 2, and ≥ 3 lines, respectively) improvement compared to baseline in mLCVA at Day 8 (excluding the primary endpoint)
Time Frame: up to 15 days
Population: miTT
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 70 | 73
Participants
  Day 8: >= 15 letters | 9 | 2
  Day 8: 10-14 letters | 20 | 14
  Day 8: 5-9 letters | 22 | 29
  Day 8: Less than 5 | 19 | 28
  Day 15: number analyzed (Participants) | 68 | 73
  Day 15: >= 15 letters | 14 | 2
  Day 15: 10-14 letters | 16 | 15
  Day 15: 5-9 letters | 28 | 39
  Day 15: Less than 5 | 10 | 17

3. Secondary Outcome: Percent of Subjects With Photopic Low Contrast Visual Acuity (pLCVA) and mHCVA Improvement in Study Eye
Description: Percent of subjects with ≥ 5, ≥ 10, and ≥ 15 ETDRS letters (≥ 1, ≥ 2, and ≥ 3 lines, respectively) improvement compared to baseline in pLCVA and mHCVA at Day 8 and Day 15
Time Frame: up to 15 days
Population: per-protocol(PP)
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 68 | 73
Participants
  pLVCA Day 8: >= 15 letters | 3 | 0
  pLVCA Day 8: 10-14 letters | 12 | 9
  pLVCA Day 8: 5-9 letters | 24 | 11
  pLVCA Day 8: Less than 5 letters | 29 | 53
  pLVCA Day 15: number analyzed (Participants) | 64 | 71
  pLVCA Day 15: >= 15 letters | 7 | 1
  pLVCA Day 15: 10-14 letters | 12 | 4
  pLVCA Day 15: 5-9 letters | 22 | 20
  pLVCA Day 15: Less than 5 letters | 23 | 46
  mHCVA Day 8: >= 15 letters | 2 | 3
  mHCVA Day 8: 10-14 letters | 5 | 3
  mHCVA Day 8: 5-9 letters | 16 | 11
  mHCVA Day 8: Less than 5 letters | 45 | 56
  mHCVA Day 15: number analyzed (Participants) | 64 | 71
  mHCVA Day 15: >= 15 letters | 3 | 5
  mHCVA Day 15: 10-14 letters | 8 | 1
  mHCVA Day 15: 5-9 letters | 19 | 14
  mHCVA Day 15: Less than 5 letters | 34 | 51

4. Secondary Outcome: Change From Baseline in Study Eye Mesopic Pupil Diameter (PD)
Description: Change from baseline in study eye mesopic PD
Time Frame: up to 15 days
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 70 | 73
millimeters
  8 Days, Change from Baseline | -1.081 (0.6931) | -0.130 (0.5608)
  15 Days, Change from Baseline | -1.083 (0.6556) | -0.121 (0.4673)

5. Secondary Outcome: Percent Change From Baseline in Study Eye Mesopic Pupil Diameter (PD)
Description: Percent change from baseline in study eye mesopic PD
Time Frame: up to 15 days
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 68 | 73
percentage of change
  8 Days, Percent Change from Baseline | -17.98 (11.542) | -2.09 (9.492)
  15 Days, Percent Change from Baseline | -18.06 (11.418) | -1.75 (7.581)

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 23/71 | 2/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phentolamine Ophthalmic Solution 0.75% (N=71) | Phentolamine Ophthalmic Solution Vehicle (N=73)
Instillation site pain (General disorders) | 9 | 0
Dysgeusia (Nervous system disorders) | 8 | 0
Conjunctival Hyperaemia (Eye disorders) | 6 | 2
Instillation site erythema (General disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT04638660/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04638660/SAP_001.pdf